CLINICAL TRIAL: NCT04495088
Title: Preoperative FOLFOX Versus Postoperative Risk-adapted Chemotherapy in Patients With Locally Advanced Rectal Cancer and Low Risk for Local Failure: A Randomized Phase III Trial of the German Rectal Cancer Study Group
Brief Title: Preoperative FOLFOX Versus Postoperative Risk-adapted Chemotherapy in Patients With Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ralf Hofheinz (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other); German Rectal Cancer Study Group (Unknown)
Responsible Party: Sponsor-Investigator, Ralf Hofheinz, Prof. Dr., Universitätsmedizin Mannheim
Organization: Universitätsmedizin Mannheim (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACO/ARO/AIO-18.2; 2018-001356-35 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy; Leucovorin; Oxaliplatin; Fluorouracil; XELOX; Adjuvants, Pharmaceutic; Capecitabine

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, two-armed
Masking Description: open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (experimental arm) (Experimental): The experimental arm A starts with 6 cycles of mFOLFOX or 4 cycles of XELOX. Surgery is scheduled four or six weeks after day 1 of the last mFOLFOX or XELOX cycle, respectively. No postoperative chemotherapy is planned
  Interventions: Drug: mFOLFOX (neoadjuvant); Drug: XELOX (neoadjuvant)
- B (control arm) (Active Comparator): In the standard arm B, patients undergo surgical resection of the primary tumor followed by stage- (risk-)adapted adjuvant chemotherapy 4-8 weeks after surgery according to recommendations of the S3 guidelines in analogy to colon cancer. Details of the recommended protocols are provided in the protocol.
  Interventions: Drug: mFOLFOX (adjuvant); Drug: XELOX (adjuvant); Drug: Capecitabine (adjuvant); Drug: infusional 5-FU/FA "AIO" regimen (adjuvant); Drug: infusional 5-FU/FA "de Gramont" (adjuvant)

INTERVENTIONS:
Drug: mFOLFOX (neoadjuvant) — neoadjuvant application Folinic acid: 400 mg/m2, 2h i.v., on day 1 Oxaliplatin: 85 mg/m2, 2-6h i.v., on day 1 5-FU: 2400 mg/m2, 46-48h i.v., on day 1. Cycles are repeated on day 15. A total of 6 cycles are administered.
  Other Names: Folinic acid, Oxaliplatin, 5-FU
  Arms: A (experimental arm)
Drug: XELOX (neoadjuvant) — neoadjuvant application Capecitabine: 1,000 mg/m2 bid, po, on days 1-14 Oxaliplatin: 130 mg/m2, 2-6h i.v. day 1 Cycles are repeated on day 22. A total of 4 cycles are administered.
  Other Names: Capecitabine, Oxaliplatin
  Arms: A (experimental arm)
Drug: mFOLFOX (adjuvant) — adjuvant application Folinic acid: 400 mg/m2, 2h i.v., on day 1 Oxaliplatin: 85 mg/m2, 2-6h i.v., on day 1 5-FU: 2400 mg/m2, 46-48h i.v., on day 1. Cycles are repeated on day 15. A total of 6 cycles are administered.
  Other Names: Folinic acid, Oxaliplatin, 5-FU
  Arms: B (control arm)
Drug: XELOX (adjuvant) — adjuvant application Capecitabine: 1,000 mg/m2 bid, po, on days 1-14 Oxaliplatin: 130 mg/m2, 2-6h i.v. day 1 Cycles are repeated on day 22. A total of 4 cycles are administered.
  Other Names: Capecitabine, Oxaliplatin
  Arms: B (control arm)
Drug: Capecitabine (adjuvant) — adjuvant application Capecitabine: 1,250 mg/m2 bid, po, on days 1-14 Cycles are repeated on day 22. A total of 8 cycles are administered.
  Other Names: Capecitabine
  Arms: B (control arm)
Drug: infusional 5-FU/FA "AIO" regimen (adjuvant) — adjuvant application Folinic acid 2h i.v. 500 mg/m² 5-FU 2,600mg/m² (24h infusion) Days 1, 8, 15, 22, 29, 36; cycle is repeated day 57 (representing one cycle); a total of 3 cycles should be administered.
  Other Names: 5-FU, Folinic acid
  Arms: B (control arm)
Drug: infusional 5-FU/FA "de Gramont" (adjuvant) — adjuvant application Folinic acid 2h i.v. 200 mg/m² days 1 and 2 5-FU 400mg/m² bolus followed by 600mg/m² 22h infusion days 1 and 2 The cycle is repeated day 15; a total of 12 cycles should be administered.
  Other Names: 5-FU, Folinic acid
  Arms: B (control arm)

SUMMARY:
This is a multicenter, prospective, randomized, stratified, controlled, open-label study comparing preoperative FOLFOX versus postoperative risk-adapted chemotherapy in patients with locally advanced rectal cancer and low risk for local failure

DETAILED DESCRIPTION:
Patients with locally advanced rectal cancer are generally treated with preoperative 5-FU- or capecitabine-based chemo-radiotherapy (CRT) and total mesorectal excision (TME) surgery in order to decrease the rate of local failure. In patients with low risk for local failure in the middle third of the rectum (cT3a/b, N-) as determined with quality controlled MRI, the German S3 guidelines and the ESMO clinical practice guidelines state that neoadjuvant radiotherapy may be omitted. However, distant failure rate is still substantial in the range of 20-25% in these patients highlighting the need for more effective systemic treatment.

The hereby proposed ACO/ARO/AIO-18.2 randomized trial incorporates three novel aspects: (1) patient selection relies on strict and quality controlled MRI features and therefore identifies a cohort without imminent need for radiotherapy, (2) the sequence of chemotherapy and surgery is changed in a way that chemotherapy is administered preoperatively to increase the rate of patients treated with chemotherapy, and (3) three months of neoadjuvant FOLFOX or XELOX (instead of up to 6 months adjuvant chemotherapy) are used as a sole perioperative treatment in order to administer effective doses of the presumably most effective perioperative treatment at an early time point during the course of disease.

Thus, patients with locally advanced rectal cancer but low risk for local failure (cT1/2N+ in all thirds of the rectum, cT3a/b N- in the middle third, and cT3-4 Nany in the upper third) will be included and randomized between three months of neoadjuvant FOLFOX/XELOX in Arm A and primary resection of the tumor followed by risk (i.e. stage) adapted chemotherapy in Arm B.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with histologically confirmed diagnosis of rectal adenocarcinoma localised 0 - 16 cm from the anocutaneous line as measured by rigid rectoscopy (i.e. lower, middle and upper third of the rectum), depending on MRI-defined inclusion criteria (see below).
2. Staging requirements: High-resolution magnetic resonance imaging (MRI) of the pelvis is the mandatory local staging procedure.
3. Transrectal endoscopic ultrasound (EUS) is used to help discriminate between T1/2 and early T3 tumors.
4. MRI-defined inclusion criteria:

   i. Lower third (0-6 cm):
   * cT1/2 with clear cN+ based on defined MRI criteria or T3a-b (i.e. maximum infiltration into the perirectal fat of 5mm), provided CRM > 2mm and EMVI-** ii. Middle third (≥ 6-12 cm):
   * cT1/2 with clear cN+ provided CRM- and EMVI-**
   * cT3 irrespective of the depth of invasion into the perirectal fat, provided no evidence that tumor is adjacent to (defined as within 2 mm of) the mesorectal fascia on MRI (i.e. CRM > 2 mm), N0 or N1, EMVI-** iii. Upper third (≥ 12-16 cm):
   * cT1/2 with clear cN+, irrespective of CRM and EMVI
   * any cT3-4 irrespective of nodal status, CRM and EMVI.
5. Spiral-CT of the abdomen and chest to exclude distant metastases.
6. Aged at least 18 years. No upper age limit.
7. WHO/ECOG Performance Status ≤1.
8. Adequate haematological, hepatic, renal and metabolic function parameters:
9. Leukocytes ≥ 3.000/mm³, ANC ≥ 2.000/mm³, platelets ≥ 100.000/mm³, Hb > 9 g/dl
10. Serum creatinine ≤ 1.5 x upper limit of normal
11. Bilirubin ≤ 2.0 mg/dl, SGOT-SGPT, and AP ≤ 3 x upper limit of normal.
12. QTc interval (Bazett**) ≤ 440 ms
13. Informed consent of the patient.

"**" Formula for QTc interval calculation (Bazett): QTc= ((QT) ̅" (ms)" )/√(RR (sec))= ((QT) ̅" (ms)" )/√(60/(frequency (1/min)))

Exclusion Criteria:

1. Distant metastases (to be excluded by CT scan of the thorax and abdomen).
2. Prior antineoplastic therapy for rectal cancer.
3. Prior radiotherapy of the pelvic region.
4. Major surgery within the last 4 weeks prior to inclusion.
5. Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
6. Subject (male or female) is not willing to use highly effective*** methods of contraception during treatment and for 6 months (male or female) after the end of treatment Male patients treated with Oxaliplatin should take legal advice concerning sperm conservation before start of therapy and should additionally use a condom during treatment period. Their female partner of childbearing potential should also use an appropriate contraceptive measure.
7. On-treatment participation in a clinical study in the period 30 days prior to inclusion.
8. Previous or current drug abuse.
9. Other concomitant antineoplastic therapy.
10. Serious concurrent diseases, including neurologic or psychiatric disorders (incl. dementia and uncontrolled seizures), active, uncontrolled infections, active, disseminated coagulation disorder.
11. Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 6 months before enrolment.
12. Chronic diarrhea (> grade 1 according NCI CTCAE).
13. Prior or concurrent malignancy ≤ 3 years prior to enrolment in study (Exception: non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1), if the patient is continuously disease-free.
14. Known allergic reactions or hypersensitivity on study medication or to any of the other excipients.
15. Evidence of peripheral sensory neuropathy > grade 1 according to CTCAE version 5.0 (see appendix).
16. Severe kidney dysfunction (creatinine clearance < 30 ml/min).
17. Recent or concurrent treatment with brivudine.
18. Pernicious or other megaloblastic anaemia caused by vitamin B12 deficiency.
19. Known dihydropyrimidine dehydrogenase deficiency.
20. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial).

"***"highly effective (i.e. failure rate of <1% per year when used consistently and correctly) methods: intravaginal and transdermal combined (estrogen and progestogen containing) hormonal contraception; injectable and implantable progestogen-only hormonal contraception; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence (complete abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | up to 3 years
  time from randomisation to one of the following events: no surgery or non-radical (R2) surgery of the primary tumour, locoregional recurrence after R0/1 resection of the primary tumour, second primary colorectal or other cancer, metastatic disease or progression, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Acute and late toxicity | From date of informed consent until the End of Treatment or 30 days after the last dose of study treatment
  assessment of acute and late toxicity according to NCI CTCAE version 5.0
Compliance (completion rate) of chemotherapy | From date of randomization until end of chemotherapy, approx. 12 (arm A) respectively up to 34 (arm B) weeks after randomization
  Rate of completion of administered chemotherapy
Surgical morbidity and complications | After surgery, approx. 2 (arm B) respectively 20 (arm A) weeks after randomization
  Surgical morbidity and complications if surgery is performed and events occur
Pathological UICC-staging, including pCR (ypT0N0) rate | After surgery, approx. 2 (arm B) respectively 20 (arm A) weeks after randomization
  Pathological staging according UICC criteria, including detailed information about pathologically assessed complete response rate (ypT0N0)
R0 resection rate, Negative circumferential resection rate (CRM > 1mm) | After surgery, approx. 2 (arm B) respectively 20 (arm A) weeks after randomization
  defined as microscopically margin negative resection with no gross or microscopic tumor remains in the area of the primary tumor and/or samples regional lymph nodes based on evaluation by the local pathologist
Tumor regression grading according to Dworak in the experimental arm | After surgery, approx. 2 (arm B) respectively 20 (arm A) weeks after randomization
  Grading of tumor regression according to Dworak in the experimental arm
Rate of sphincter-sparing surgery | After surgery, approx. 2 (arm B) respectively 20 (arm A) weeks after randomization
  Rate of sphincter-sparing surgery if surgery is performed
Rate of W&W with or without local regrowth | Up to 5 years after end of treatment
  Number of performed watch&wait approaches with or without local regrowth compared to planned and performed surgery
Cumulative incidence of local and distant recurrences | Up to 5 years after end of treatment
  Total number of local and distant recurrences, if they occur
Overall survival | Up to at least 3 years and until 5 years
  Overall survival is defined as the time interval between the date of randomization and the date of death of any cause. Patients who are still alive when last traced will be censored at the date of last follow-up
Patient reported outcome: Quality of life according to questionnaire EORTC-QLQ-C30 | From date of randomization until the date of first documented progression or date of death from any cause, whichever occured first, assessed up to approximately 68 months
  Quality of life scores according to validated questionnaires EORTC-QLQ-C30, based on treatment arm, and surgical procedures. 30 questions; score values from 1 (not at all) to 4 (very much) respectively from 1 (very poor) to 7 (excellent). Score outcome depends on score type.
Patient reported outcome: Quality of life according to questionnaire EORTC-QLQ-CR29 | From date of randomization until the date of first documented progression or date of death from any cause, whichever occured first, assessed up to approximately 68 months
  Quality of life scores according to validated questionnaires EORTC-QLQ-CR29, based on treatment arm, and surgical procedures. 29 questions; score values from 1 (not at all) to 4 (very much). Score outcome depends on score type.
Patient reported outcome: Functional outcome according to Wexner score | From date of randomization until the date of first documented progression or date of death from any cause, whichever occured first, assessed up to approximately 68 months
  Functional score according to validated Wexner score, based on treatment arm, and surgical procedures. 5 questions; five score values from "never" to "1 per day or more often". The more often the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf-Dieter Hofheinz, Prof. Dr., Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Unversity Hospital Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No